CLINICAL TRIAL: NCT04063462
Title: A Phase 2 Study of Pyrotinib in Patients With Non-Small Cell Lung Cancer (NSCLC), With at Least One Prior Systemic Treatment, Locally Advanced or Metastatic, With EGFR or ERBB2 Exon 20 Insertion Mutation (PEER20)
Brief Title: Phase 2 Study of Pyrotinib in Previously Treated Patients With NSCLC Having EGFR or ERBB2 Exon 20 Insertion Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEER20
Record Dates: First submitted 2019-07-21; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Previously treated patients with EGFR exon 20 insertion mutant positive NSCLC
  Interventions: Drug: Pyrotinib
- Cohort 2 (Experimental): Previously treated patients with HER2 exon 20 insertion mutant positive NSCLC
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — pyrotinib, single agent, 400mg p.o once daily until disease progressed

SUMMARY:
This is a Phase 2, open-label study to evaluate the efficacy and the safety/tolerability of pyrotinib in previously treated NSCLC patients with EGFR exon 20 insertion mutations or HER2 exon 20 insertion mutations. Patient has had at least one prior systemic treatment for locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80years，ECOG PS：0-2，Life expectancy of more than 3 months，with measurable lesion ( RECIST1.1).
2. Histologically or cytologic confirmed EGFR or HER2 Exon 20 Insertion Mutation positive advanced Non-small cell lung cancer who failed prior therapies.
3. ≥1 target lesion that has not received radiotherapy in the past 3 months and can be accurately measured in at least 1 direction；Previously received radiation therapy, but the radiotherapy area must be <25% of the bone marrow area, and radiation therapy must have closed for at least≥4 weeks at the time of enrollment.
4. Main organs function is normal.
5. Signed and dated informed consent.

Exclusion Criteria:

1. Patient has had previous treatment with Pyrotinib, Poziotinib or any other EGFR or HER2 exon 20 insertion mutation-selective tyrosine kinase inhibitor (TKI) prior to study participation. The currently approved TKIs (ie, erlotinib, gefitinib, afatinib, osimertinib) are not considered to be exon 20 insertion-selective and are permissible
2. Patients who planned to receive systemic anti-tumor therapy within 4 weeks prior to allocation or during the course of this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or receiving the Mitomycin C 6 weeks prior to medication). Extra-field radiotherapy (EF-RT) was performed 4 weeks prior to allocation or restricted radiotherapy for assessing tumor lesions within 2 weeks prior to allocation
3. With kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus)
4. Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pyrotinib
6. History of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplantation; active infection including hepatitis B (HBV DNA level ≥1000 copies /mL), hepatitis C and human immunodeficiency virus (HIV); Severe acute or chronic infections requiring systemic treatment
7. Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial
8. Known history of neurological or psychiatric disease, including epilepsy or dementia
9. Has a history of malignant tumors. Except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone curative treatment and have no disease recurrence within 5 years after the start of treatment
10. Respiratory syndrome (dyspnea≥CTC AE 2), severe pleural effusion, ascites, pericardial effusion
11. Abnormal blood coagulation (INR>1.5 or PT > ULN + 4s or APTT > 1.5 ULN), with bleeding tendency or receiving thrombolytic or anticoagulant therapy; Renal insufficiency: urinary protein ≥ ++, or 24-hour urine protein ≥ 1.0g
12. Patient has had other malignancies within the past 3 years, except for stable non-melanoma skin cancer, fully treated and stable early stage prostate cancer or carcinoma in situ of the cervix or breast without need of treatment
13. Patient is pregnant or breast-feeding
14. Judgment by the investigator that should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | To evaluate objective response rate 6-8 weeks after the initiation of pyrotinib
  The proportion of subjects who achieve Complete Response (CR) and Partial Response (PR) by the best response from the first dose of pyrotinib to the end of study.

SECONDARY OUTCOMES:
Progression Free Survival | 24 months
  The PFS time is defined as time from enrollment to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of : "death", "last tumor assessment", "last follow up date" or "last date in drug log"
Disease Control Rate (DCR) | 24 months
  Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
OS（Overall Survival） | 24 months
  OS was defined as time from date of enrollment to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
Duration of Response (DoR) | 24 months
  Number of days from the date that measurement criteria are first met for CR or PR (whichever status is recorded first) until the first subsequent date that progressive disease or death is documented.
Safety and Tolerability | 24 months
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individul participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requestors will be required to sign a Data Access Agreement.